CLINICAL TRIAL: NCT03359148
Title: Potential Risk for Bacterial Contamination in Conventional Reused Ventilator Systems and Disposable Closed Ventilator-Suction Systems
Brief Title: Potential Risk for Bacterial Contamination in Ventilator Systems
Status: Completed | Type: Observational
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Gwo-Hwa Wan, Professor, Chang Gung University
Other Study IDs: CMRPD1D0251
Record Dates: First submitted 2017-11-21; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Contaminated Medical or Biological Substances; Environmental-Pollution-Related Condition
Keywords: Nosocomial infection; Ventilator system; Closed suction system; Open suction system; Bacterial contamination
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disposable ventilator system: The experimental study group will be assigned to a disposable ventilator system combined with an auto-filled heated humidifier (HH), a closed suction catheter, and a closed aerosol therapy procedure with a valved T-adaptor.
  Interventions: Device: Disposable ventilator system
- Conventional reused ventilator system: According to clinical commonly used system, the control study group will be assigned to use with conventional reused ventilator system, combined with a manually filled HH, an open suction catheter, and a conventional aerosol therapy procedure.
  Interventions: Device: Conventional reused ventilator system

INTERVENTIONS:
Device: Disposable ventilator system
  Groups: Disposable ventilator system
Device: Conventional reused ventilator system
  Groups: Conventional reused ventilator system

SUMMARY:
Background: Few studies have investigated the difference of bacterial contamination between conventional reused ventilator systems and disposable closed ventilator-suction systems. The aim of this study was to investigate the bacterial contamination rates of the reused and disposable ventilation systems, and the association between system disconnection and bacterial contamination of ventilator systems.

Methods: The enrolled patients used a conventional reused ventilator system and a disposable closed ventilator-suction system, respectively, for a week; specimens were then collected from the ventilators' internal system to evaluate human and environmental bacterial contamination. The sputum specimens from patients were also analyzed in this study.

Results: The detection rate of bacteria in the conventional reused ventilator system was substantially higher than that in the disposable system. The inspiratory and expiratory limbs of disposable closed ventilator-suction system had higher bacterial concentrations than the conventional reused ventilator system. The bacterial concentration in the heated humidifier (HH) of the reused system was significantly higher than that in the disposable system. Positive associations existed among the bacterial concentrations at different locations in the reused and disposable ventilator systems, respectively. The predominant bacteria identified in the reused and disposable ventilator systems included Acinetobacter spp., Bacillus cereus, Elizabethkingia spp., Pseudomonas spp., and Stenotrophomonas (Xan) maltophilia.

Conclusion: Both the reused and disposable ventilation systems had high bacterial contamination rates after one week of use. Disconnection of the ventilator systems should be avoided during system operation for decreasing the risks of environmental pollution and human exposure, especially for the disposable system.

DETAILED DESCRIPTION:
The intubated and mechanically ventilated patients were enrolled from the Intensive Care Unit of Chang Gung Memorial Hospital, Taiwan. The experimental study group was assigned to a disposable ventilator system combined with an auto-filled heated humidifier (HH), a closed suction catheter, and a closed aerosol therapy procedure with a valved T-adaptor. According to clinical commonly used system, the control study group was assigned to use with conventional reused ventilator system, combined with a manually filled HH, an open suction catheter, and a conventional aerosol therapy procedure. Every patient was use above both ventilator systems.

ELIGIBILITY:
Inclusion Criteria:

* the mechanically ventilated patients in the ICU

Exclusion Criteria:

* the sputum culture results of the patients indicated the presence of drug-resistant bacteria, influenza virus, and early extubation.

Ages: 20 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 16 patients (10 men and 6 women, aged between 20 and 91 years) were included for the final analysis. Patients had been on a mechanical ventilator for 17-46 days, and had a primary diagnosis of sepsis, septic shock, cardiac arrest, pneumonia (CAP or HAP), chronic obstructive pulmonary disease, respiratory failure, acute respiratory distress syndrome, or lung contusion.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
bacterial concentration | 7 days later
  comparison of the two ventilator systems

SECONDARY OUTCOMES:
bacterial detection rate | 7 days later
  comparison of the two ventilator systems

CONTACTS AND LOCATIONS:
Overall Officials: GWO-HWA WAN, Ph.D., Principal Investigator — Chang Gung University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li YC, Lin HL, Liao FC, Wang SS, Chang HC, Hsu HF, Chen SH, Wan GH. Potential risk for bacterial contamination in conventional reused ventilator systems and disposable closed ventilator-suction systems. PLoS One. 2018 Mar 16;13(3):e0194246. doi: 10.1371/journal.pone.0194246. eCollection 2018. PMID 29547638